CLINICAL TRIAL: NCT07269041
Title: A Phase I Feasibility Study of HSPC Infusion Following Total Lymphoid Irradiation and Anti-thymocyte Globulin in Patients With a Pre-existing, Well-functioning HLA-matched Living-donor Liver Transplant to Induce Immune Tolerance.
Brief Title: Immune Tolerance Induction After Liver Transplantation
Acronym: iTILT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Cray V. Noah, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25-2369
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplantation; Immune Tolerance; Immune Tolerance/Drug Effects; Graft Survival; Hematopoietic Stem Cell; Chimerism; Immunosuppression After Liver Transplantation; Immunosuppression Disorders; End Stage Liver Disease
Keywords: Liver Transplantation; Immune Tolerance; Hematopoietic Stem Cell Infusion; Chimerism; Mixed Chimerism; Total Lymphoid Irradiation; Antithymocyte Globulin; Immunosuppression Withdrawal; Living Donor Liver Transplant; Tolerance Induction; Delayed Immune Tolerance; Retroactive Immune Tolerance; Immunosuppression Toxicity
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tolerance Induction Arm (Experimental): Adult recipients with a pre-existing, well-functioning HLA-matched living-donor liver transplant from the same donor will undergo outpatient conditioning with total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (rATG), followed by infusion of mobilized donor hematopoietic stem and progenitor cells (separate CD34+ and CD3+ fractions). After HSPC infusion, participants will be monitored for donor chimerism, graft function, rejection, and GVHD, and will undergo a structured taper of maintenance immunosuppression with the goal of complete withdrawal if donor chimerism is present and protocol criteria are met.
  Interventions: Biological: Donor Hematopoietic Stem and Progenitor Cell Infusion

INTERVENTIONS:
Biological: Donor Hematopoietic Stem and Progenitor Cell Infusion — Participants with a pre-existing, well-functioning HLA-matched living-donor liver transplant from the same donor will receive a delayed infusion of donor-derived hematopoietic stem and progenitor cells (HSPCs). Donors undergo mobilization and apheresis to collect peripheral blood stem cells, which are processed to generate a CD34+ cell product with an accompanying defined CD3+ T-cell dose. Recipients receive outpatient conditioning with total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (rATG) prior to infusion. The goal of the intervention is to induce tolerance by achieving durable mixed chimerism and enable structured withdrawal of maintenance immunosuppression.
  Other Names: Donor HSPC Infusion

SUMMARY:
This clinical trial is being conducted to help liver transplant recipients safely discontinue toxic immunosuppressive drugs years after surgery. Lifelong use of these drugs is the current standard, but they come with life-threatening side effects. UCLA has pioneered this "Delayed Tolerance" approach, achieving success in numerous kidney recipients now living drug-free. The process uses a conditioning regimen followed by donor stem cell infusion to retrain the immune system to accept the liver as "self."

DETAILED DESCRIPTION:
This study seeks to determine if patients with a pre-existing, well-functioning liver transplant from an HLA-matched living donor can be withdrawn from maintenance immunosuppressive medications without compromising allograft function through hematopoietic stem and progenitor cell (HSPC) infusion from the same donor. HSPC infusion will be preceded by a conditioning regimen of total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (rATG) that takes course over two weeks, with HSPC infusion being on the final day. This entire protocol will take place in the outpatient setting.

At serial time points, (1) graft function will be monitored, (2) chimerism will be measured in recipient whole blood and white blood cell subsets, and (3) protocol biopsies of the graft will be obtained. An attempt will be made to discontinue tacrolimus. Weaning of tacrolimus will begin at 6 months with a goal of discontinuation by 10-12 months as long as the following conditions are met: (1) donor chimerism is detectable for at least 180 days after HSPC infusion, (2) stable graft function (defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and total bilirubin (TBil) levels each ≤ 2.0 × the upper limit of normal) is maintained without clinical or biopsy-determined rejection episodes, and (3) there is no evidence of graft-versus-host disease . HSPC infusion will consist of a target dose of 10 x106 CD34+ cells/kg and 5 x106 CD3+ cells/kg with the goal of achieving durable mixed chimerism.

Immunological tolerance through combined solid organ and HSPC transplant has been demonstrated at a few centers of excellence within the United States, including UCLA. The aim of these protocols is to liberate patients from lifelong immunosuppression. Thus far, protocols have been largely limited to HLA-matched donor recipient pairs undergoing simultaneous kidney and HSPC transplant from the same donor. In all protocols, the recipient undergoes a conditioning regimen to facilitate HSPC engraftment. At UCLA, our protocol employs a conditioning regimen of TLI and ATG. We are the first center to demonstrate the feasibility of retroactive immune tolerance, where a patient with a pre-existing fully HLA-matched kidney transplant underwent HSPC infusion following a conditioning regimen of TLI and ATG over one year after the kidney transplant surgery and successfully achieved durable mixed chimerism and tolerance, allowing permanent discontinuation of immunosuppressants - a process called "delayed tolerance."

Though the liver has intrinsic tolerogenic properties, tolerance protocols for liver are largely limited by the medical and logistical demands of recovering from liver transplant. As we have demonstrated in our single center experience, delayed tolerance has potential to be a reproducible strategy to permanently discontinue immunosuppressants in recipients who receive HSPC transplant months to years after transplant surgery. As such, recipients of HLA-matched living-donor liver transplants who have recovered from their surgery may benefit from protocols to establish tolerance and liberate them from lifelong immunosuppression.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Males and females ages 18 years and older with a pre-existing liver transplant from a living donor with a donor-recipient match at 6 or more out of 12 alleles across the HLA-A, -B, -C, -DR, -DQ, and -DP loci, as determined by high-resolution HLA typing.
2. Pre-existing living-donor liver transplant must be 12 months to 20 years from date of scheduled HSPC infusion.
3. Agreement to participate in the study and ability to give informed consent.
4. Liver biopsy within 4 weeks of enrollment without signs of rejection.
5. Meets institutional criteria for HSPC infusion.
6. Resides or is willing to stay within 3 hours distance from UCLA Medical Center by ground transportation for the first three months of the trial at the physician's discretion.
7. No known contraindication to administration of rATG or radiation therapy.
8. If subject is a female of reproductive potential (i.e., no documented absence of ovaries or uterus, history of tubal ligation, or post-menopausal status), subject must be confirmed not pregnant by a serum or urine pregnancy test and must agree to practice a reliable form of contraception including hormonal treatments, barrier methods or intrauterine device for at least 12 months following initiation of the tolerance protocol.

Recipient Exclusion Criteria:

1. Major ABO incompatibility with donor.
2. Any of the following labs > 2.0 times the upper limit of normal on screening: AST, ALT, ALP, GGT or TBil.
3. History of rejection with current HLA-matched liver transplant within the last year.
4. History of GVHD following liver transplant.
5. Positive Class II HLA Donor-Specific Antibody (DSA) or class I DSA specificity above 5,000 MFI at the time of the stem cell infusion.
6. History of multi-organ transplantation, either simultaneous or as separate events.
7. History of more than one liver transplant.
8. Known allergy to rabbit proteins.
9. History of a major post-transplant complication at investigator discretion.
10. History of active malignancy within the past 5 years except for:

    1. Malignancy that has not required treatment in the past on active surveillance.
    2. Malignancy treated with curative intent with no known active disease >2 years before the first dose of study treatment and of low potential risk for recurrence.
    3. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    4. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ, DCIS).
11. Active bacterial, fungal or mycobacterial infection.
12. Clinically significant viremia from EBV, CMV, HCV or HBV PCR test within the past 3 months.

    1. Significant CMV viremia is defined as greater than or equal to 137 IU/mL.
    2. If CMV low-level viremia is detected, defined as 137 - 1,000 IU/mL, patients may undergo subsequent testing up to twice per week and two consecutive negative results will allow for inclusion.
13. Seropositivity for HIV 1 or 2 by 4th generation serum antibody/antigen testing, or HTLV I or II by serum antibody testing.
14. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
15. Active extra-hepatic autoimmune disease requiring immunosuppression.
16. Autoimmune disease was the indication for liver transplantation.
17. Any condition that precludes the ability to give informed consent and/or places the subject at high risk for non-compliance with the safety monitoring requirements of the study.
18. Received immunotherapy drugs, such as immune checkpoint inhibitors (e.g. pembrolizumab, nivolumab, and ipilimumab), tumor necrosis factor inhibitors, rituximab, or interleukin-2 within six months of the study treatment.
19. Use of medications with known hepatotoxicity or potential to confound interpretation of liver function tests (e.g., methotrexate, isoniazid, amiodarone), unless reviewed and approved by the Principal Investigator and hepatology, and the subject has demonstrated stable liver function tests for ≥6 months while on the medication.
20. Active hepatobiliary and pancreatic diseases:

    1. History of chronic hepatobiliary or pancreatic disorders that may interfere with safety assessments or interpretation of protocol endpoints, including but not limited to primary sclerosing cholangitis (PSC), autoimmune hepatitis, primary biliary cholangitis (PBC), chronic pancreatitis, recurrent cholangitis, biliary strictures, biliary obstruction, untreated bile duct injury, hepatobiliary malignancy, or metabolic/genetic liver disease (e.g., Wilson's disease, alpha-1 antitrypsin deficiency).
    2. Active chronic liver diseases such as metabolic dysfunction-associated steatohepatitis (MASH) and alcohol-associated liver disease.
    3. Gallbladder diseases such as cholecystitis or symptomatic cholelithiasis.

Donor Inclusion Criteria:

1. Males and females ages 18 years and older meeting the HLA-matching requirements specified in the "Recipient Inclusion Criteria" above.
2. Must meet the following criteria for HSPC donation:

   1. Hgb: > 11 g/dl
   2. Plt: > 80,000/µL
   3. WBC: > 3,000/µL

Donor exclusion criteria:

1. Major ABO incompatibility with recipient.
2. Medically unfit to tolerate peripheral blood apheresis (e.g., small body size, poor vascular access, not a suitable candidate for placement of a central catheter).
3. Pregnant (confirmed by urine or serum pregnancy test) or lactating.
4. Seropositivity for HIV 1 or 2 by 4th generation serum antibody/antigen testing, HTLV I or II by serum antibody testing.
5. Active West Nile Virus infection.
6. Active bacterial, fungal, mycobacterial or viral infection (including active hepatitis B and/or C).
7. Psychiatric, addictive, neurological, or other disorder that compromises ability to give true informed consent for participation in this study
8. Use of oral anticoagulants within two days of apheresis.
9. History of active malignancy within the past 5 years except for:

   1. Malignancy that has not required treatment in the past on active surveillance.
   2. Malignancy treated with curative intent with no known active disease >2 years before the first dose of study treatment and of low potential risk for recurrence.
   3. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   4. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ, DCIS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects weaned off liver transplant immunosuppressants at 12 months after HSPC infusion | 12 months post-HSPC infusion.
  The percentage of subjects who successfully discontinue all liver transplant immunosuppressant medications at 12 months after HSPC infusion.

SECONDARY OUTCOMES:
Liver graft rejection within 48 months post-HSPC infusion | Up to 48 months post-HSPC infusion.
  Percentage of subjects with liver graft rejection within 48 months after HSPC infusion, defined as:
  1. meeting Banff criteria for rejection on biopsy obtained to confirm clinical suspicion, or
  2. clinical suspicion of rejection with response to corticosteroids when biopsy is contraindicated or declined.
Graft failure | Up to 48 months post-HSPC infusion.
  Percentage of subjects with graft failure as determined by re-listing for liver transplantation and/or re-transplantation.
Incidence of GVHD | Up to 48 months post-HSPC infusion.
  Incidence of graft-versus-host disease (GVHD) defined as grade ≥2 acute GVHD or score ≥2 chronic GVHD.

OTHER OUTCOMES:
Chimerism persistence | 12, 24, 36, and 48 months post-HSPC infusion.
  Percentage of subjects with detectable donor-recipient chimerism for at least 180 days within the first 12 months after HSPC infusion, and at 12, 24, 36, and 48 months.
Incidence of acute or chronic GVHD (detailed) | Up to 48 months post-HSPC infusion
  Percentage of subjects that experienced acute or chronic GVHD, diagnosed clinically and/or by biopsy of the affected organ.
Liver function | 12, 24, 36, and 48 months post-HSPC infusion.
  Percentage of subjects with normal liver function tests (AST, ALT, ALP, TBil, and GGT each ≤ 2× upper limit of normal) at 12, 24, 36, and 48 months.
Infection burden | 12, 24, 36, and 48 months post-HSPC infusion.
  Mean number of bacterial, fungal, and viral infections per subject at 12, 24, 36, and 48 months.
Change in medication use for metabolic syndrome | 6, 12, 24, 36, and 48 months post-HSPC infusion.
  Percentage and average change in dosing of subjects requiring medications for hypertension, diabetes, and hyperlipidemia at Months 6, 12, 24, 36, and 48.
Quality of Life as Assessed by Change from Baseline in PROMIS-29 Profile v2.1 Through Month 48 | Baseline, Day 14, and Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 18, 24, 36, and 48 post-HSPC infusion
  The Patient-Reported Outcomes Measurement Information System 29-Item Profile v2.1 (PROMIS-29 Profile v2.1) is a validated 29-item patient-reported outcome measure assessing physical, mental, and social health in liver transplant recipients. Domains include physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and social roles.
Quality of Life as Assessed by Change from Baseline in MTSOSD-R 59 Through Month 48 | Baseline, Day 14, and Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 24, 36, and 48 post-HSPC infusion
  Modified Transplant Symptom Occurrence and Symptom Distress Scale - Revised (MTSOSD-R 59) is a transplant-specific symptom inventory that assesses symptom occurrence and associated distress in immunosuppressed liver transplant recipients across multiple domains.
Quality of Life as Assessed by Change from Baseline in pLTQ Through Month 48 | Baseline, and Months 6, 12, 24, 36, and 48 post-HSPC infusion
  Post-Liver Transplant Quality of Life Instrument (pLTQ) is a liver transplant-specific quality-of-life instrument assessing physical, psychological, and social functioning domains relevant to long-term transplant outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Veale, MD, Principal Investigator — UCLA Health; Cray V. Noah, MD, Study Director — UCLA Health
Locations (1):
- UCLA Health 200 Medical Plaza, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because this is a Phase I, single-site study involving transplant recipients and their living donors, where data elements such as HLA high-resolution typing, chimerism profiles, and longitudinal graft function measurements are inherently identifiable. Sharing raw IPD would pose a significant re-identification risk and is not permitted under the study's IND, IRB approval, or institutional policies for early-phase cellular therapy trials. Aggregate, de-identified results will be disseminated through scientific publications and presentations, but participant-level datasets will not be made publicly available.

REFERENCES:
- [Background] Nassiri N, Lum E, Mead MD, Raldow AC, Kogut N, Veale JL. Immune tolerance induction through haematopoietic chimerism after kidney donation. Lancet. 2022 Aug 6;400(10350):e2. doi: 10.1016/S0140-6736(22)00914-X. No abstract available. PMID 35934008
- [Background] Lum EL, Nassiri N, Kogut N, Oliai C, Raldow A, Reed EF, Veale JL. Delayed immune tolerance through donor haematopoietic stem cell infusion 14 months after kidney transplantation. Lancet. 2024 Oct 5;404(10460):1346. doi: 10.1016/S0140-6736(24)01935-4. No abstract available. PMID 39368842
- See also: UCLA Immune Tolerance Website — https://www.uclahealth.org/medical-services/transplants/kidney-transplant/living-donor-transplant/immunosuppression-free-kidney-transplant-tolerance-program